CLINICAL TRIAL: NCT06334055
Title: Validation Study of Mean Arterial Pressure (MAP) Parameter of Masimo INVSENSOR00073
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1091
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo INVSENSOR00073 sensor.
  Interventions: Device: Masimo INVSENSOR00073

INTERVENTIONS:
Device: Masimo INVSENSOR00073 — Noninvasive blood pressure monitor

SUMMARY:
The aim of the study is to validate the Mean Arterial Pressure (MAP) parameter of Masimo INVSENSOR00073 against the gold standard blood pressure measurements from the arterial line while subject undergo a blood pressure variation procedure.

ELIGIBILITY:
Inclusion Criteria:

Influenced by study design:

* Subject is 18 to 40 years of age.
* Subject weighs a minimum of 110 lbs.
* Baseline heart rate ≥ 45 bpm and ≤ 90 bpm.
* Baseline blood pressure:
* Systolic blood pressure ≤ 135 mmHg and ≥ 100 mmHg.
* Diastolic blood pressure ≤ 95 mmHg and ≥ 55 mmHg.
* Valid systolic blood pressure (SBP) auscultatory measurements for lateral difference is ≤ 15 mmHg.
* Valid diastolic blood pressure (DBP) auscultatory measurements for lateral difference is ≤ 10 mmHg.
* Hemoglobin value ≥ 11 g/dL.
* CO value ≤ 3.0% FCOHb.
* Subject is comfortable to read and communicate in English*. * This is to ensure the subject can provide informed consent (as study materials are currently available in English only) and can comply with study procedures.

Exclusion Criteria:

Influenced by device warning labels:

* Subject is pregnant or breastfeeding.
* Subject is experiencing dysrhythmia or arrhythmia.

Influenced by study design/environment:

* Subject is concurrently participating in another research study.
* Subjects not suitable for the investigation at the discretion of the clinical team including but not limited to the items below.
* Subjects who do not pass the health assessment for safe participation in the study procedures.
* Inability to insert or difficulty with inserting an intravenous line in the subject's hand or arm and/or an arterial line in the radial artery of the subject's wrist.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Masimo INVSENSOR00073: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo INVSENSOR00073 sensor.
  Masimo INVSENSOR00073: Noninvasive blood pressure monitor
Period: Overall Study
Arm/Group | Masimo INVSENSOR00073
Started | 101
Completed | 25
Not Completed | 76
Not completed — Adverse Event | 4
Not completed — Disqualified | 72

BASELINE CHARACTERISTICS:
Arm/Group | Test Subject
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure (MAP) Accuracy and Precision of Masimo INVSENSOR00073
Description: Accuracy and precision of mean arterial pressure (MAP) measured by Masimo INVSENSOR00073 in comparison to radial arterial line.
Time Frame: 1-5 hours.
Population: 9 subjects not analyzed due to incorrect software version
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Masimo INVSENSOR00073
Number analyzed (Participants) | 16
Millimeters of mercury (mmHg) | 1.38 (4.98)

ADVERSE EVENTS:
Time Frame: 1-5 hours
Arm/Group | Masimo INVSENSOR00073
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 10/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Masimo INVSENSOR00073 (N=101)
Venous sample complications (Injury, poisoning and procedural complications) | 4
Arterial line complications (Injury, poisoning and procedural complications) | 2
Infusion effects (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT06334055/Prot_SAP_000.pdf